CLINICAL TRIAL: NCT03179007
Title: A Clinical Study of CTLA-4 and PD-1 Antibodies Expressing MUC1-CAR-T Cells for Patients With MUC1 Positive Advanced Solid Tumors
Brief Title: CTLA-4 and PD-1 Antibodies Expressing MUC1-CAR-T Cells for MUC1 Positive Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Cell Therapy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2017-04-P01
Record Dates: First submitted 2017-06-05; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Advanced Solid Tumor
Keywords: MUC1; CTLA-4; PD-1; chimeric antigen receptor T cells; solid tumor
MeSH Terms: conditions — Diabetes Mellitus, Insulin-Dependent, 12 | interventions — CTLA-4 Antigen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CTLA-4/PD-1 expressing MUC1-CAR-T (Experimental): This study have only one arm that is anti-CTLA-4/PD-1 expressing MUC1-CAR-T group. All patients with advanced solid tumor will take part in the screening, who matching all the conditions will be chosen for the treatment using CTLA-4 and PD-1 antibodies expressing MUC1-targeted CAR-T cells. New CAR-T cells are cultured from PBMC and returned to the patients by venous transfusion.
  Interventions: Biological: Anti-CTLA-4/PD-1 expressing MUC1-CAR-T

INTERVENTIONS:
Biological: Anti-CTLA-4/PD-1 expressing MUC1-CAR-T — Every cycle, peripheral blood mononuclear cells (PBMC) are collected on day 0, CAR-T cells are cultured in a GMP standard workshop. Patients are given a three-day regimen of chemotherapy consisting of cyclophosphamide aimed to deplete the lymphocytes before cells infusion. Then the patients will receive an i.v.gtt infusion of CTLA-4 and PD-1 antibodies expressing MUC1 targeted CAR-T cells at (2-5) ×10^7 cells/kg from day 18 to day 19 (±2 days). 2 cycles are regarded as a treatment period.
  Other Names: CTLA-4 and PD-1 antibodies expressing MUC1-CAR-T cells

SUMMARY:
This is a single-arm, open-label, one center clinical study, to determine the safety and efficacy of infusion of autologous T cells engineered to express immune checkpoint antibodies (CTLA-4 and PD-1) and chimeric antigen receptor targeting MUC1 in adult patients with MUC1 positive, advanced recurrent or refractory malignant solid tumors.

DETAILED DESCRIPTION:
This study will be conducted using a phase I/II trial design to assess the safety and efficacy of the CTLA-4 and PD-1 antibodies expressing MUC1-CAR-T for patients with MUC1 positive, advanced recurrent or refractory malignant solid tumors. MUC1-CAR-T can specificly and effectively kill the MUC1 positive cancer cells, CTLA4 and PD-1 antibodies are secreted from the CAR-T cells could improve immunosuppression microenvironment, new CAR-T cells contain the advantages of CAR-T and immune checkpoint inhibitor, which is a promising therapeutic method for advanced solid tumors.

The new CAR-T therapy is applied to clinical practice as bellow. T cells are prepared from peripheral blood mononuclear cells (PBMC) by leukapheresis, and then activated and engineered to express CTLA-4 and PD-1 antibodies and chimeric antigen receptor targeting MUC1. Cells are proliferated in culture and returned to the patients by venous transfusion. A total of 40 patients may be enrolled in the study. The total duration of the study is expected to be approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with relapsed or refractory advanced solid malignancies (diagnosed by histology or cytology detection).
2. Progressive disease and no response after at least second-line therapy.
3. Gender unlimited, age from 18 years to 80 years.
4. Life expectancy≥3 months.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
6. Adequate venous access for peripheral blood mononuclear cell (PBMC) apheresis, and no other contraindications.
7. Immunohistochemistry (IHC) score of MUC1 on tumor tissue ≥1+.
8. Adequate hepatic function, renal function and bone marrow function (withhin 7 days before enrollment): white blood cell (WBC)≥3.0×10^9/L; platelet≥100×10^9/L; hemoglobin≥90 g/L; lymphocyte ≥0.7×10^9/L; total bilirubin ≤2 times the upper limit of the normal value; alanine aminotransferase and aspartate transaminase (ALT and AST) ≤2.5 times the upper limit of the normal value; serum creatinine ≤1.5 times the upper limit of the normal value.
9. There is no other treatments (chemotherapy, radiotherapy, etc.) within four weeks before enrollment.
10. There is at least one measurable tumor lesion.
11. Patients have adequate ability to understand, sign informed consents and take part in the clinical research voluntarily.
12. Female patients in child bearing period must have evidence of negative pregnancy test, and agree to take effective contraceptive measures until 4 months after cells infusion.

Exclusion Criteria:

1. Patients with two or more kinds of tumors.
2. Patients with active viral or bacterial infection, and have failed to be controlled by anti-infective treatment.
3. Patients with seropositive reponse of Human immunodeficiency virus (HIV) and syphilis, or fail to control the hepatitis B virus or hepatitis C virus infection.
4. Patients with active rheumatic diseases, organ transplantation and other diseases affecting the immune system seriously.
5. Patients with severe heart and lung dysfunction.
6. Patients with severe chronic diseases of kidney, liver and other important organs.
7. Patients with any other serious illnesse that the investigators consider it will may affect the patient's treatments, follow-up or assessment, including any uncontrolled clinically significant neurological or psychiatric disorders, immunoregulatory diseases, metabolic diseases, infectious diseases and so on.
8. Patients who take part in clinical trials of other drugs or biological therapy at present or within 30 days before enrollment.
9. Patients who need long-term use of immunosuppressive drugs or patients who are undergoing treatment of autoimmune diseases.
10. Patients who need long-term use of glucocorticoid.
11. Women patients in gestation period or suckling period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-06-07 (Estimated); Primary Completion 2019-01-20 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
Safety of infusion of autologous CTLA-4 and PD-1 antibodies expressing MUC1-targeted CAR-T cells | 2 years
  Determine the toxicity profile of CTLA4 and PD-1 antibodies expressing MUC1-targeted CAR-T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
The efficacy of the treatment using CTLA-4 and PD-1 antibodies expressing MUC1-CAR-T cells for advanced solid tumors | 2 years
  The efficacy of the treatment is assessed according to the response evaluation criteria in solid tumor version 1.1 (RECIST1.1), which is defined as complete remission (CR), partial remission (PR), stable disease (SD), or progressive disease (PD).

OTHER OUTCOMES:
Progression free survival | 2 years
  Progression free survival is defined as the time from the day in which the patient is enrolled to the date on which tumor progresses or the date on which the patient dies for any cause.
Overall survival | 2 years
  Overall survival is defined as the time from the day in which the patient is enrolled to the date on which the patient dies for any cause.
Change of life quality | 2 years
  Life quality is assessed before and after the treatment.
Proliferation and persistence of MUC1 specific CAR-T cells in peripheral blood of the patients after treatment | 6 months
  CAR-T proportion in peripheral blood of the patients is detected by flow cytometry assay to study the proliferation and persistence of MUC1 specific CAR-T cells.
CTLA-4 and PD-1 antibodies level in peripheral blood of the patients after treatment | 6 months
  CTLA-4 and PD-1 antibodies level are detected by ELISA assay to asess the expressing level of CTLA4 and PD-1 antibodies from CAR-T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Qijun Qian, Ph.D, Study Chair — Shanghai Cell Therapy Research Institute; Huajun Jin, Ph.D, Study Chair — Shanghai Cell Therapy Research Institute; Zhiwei Zhang, Ph.D, Study Director — Shanghai Cell Therapy Research Institute; Yan Sun, Study Director — Shanghai Cell Therapy Research Institute; Jiangtao Wang, Principal Investigator — Ningbo No.5 Hospital(Ningbo Cancer Hospital)
Locations (1):
- Ningbo No.5 Hospital (Ningbo Cancer Hospital), Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No